CLINICAL TRIAL: NCT06678477
Title: Comparison of the Performance Between Conventional Colonoscopy and 3D Colonoscopy in Positive Fecal Immunochemical Test Group: a Multi-center, Randomized Controlled Trial
Brief Title: Comparison of the Performance Between Conventional Colonoscopy and 3D Colonoscopy in Positive Fecal Immunochemical Test Group
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, Statistical Center, NTUHCTC, Dr., National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 202311028DIPA
Record Dates: First submitted 2024-11-06; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Adenoma Detection Rate; Colonoscopy; Three Dimensional; Fecal Immunochemical Test
Keywords: colonoscopy; adenoma detection rate; 3D; Fecal immunochemical test

STUDY DESIGN:
Intervention Model Description: 3D colonoscopy versus standard 2D colonoscopy in positive FIT groups
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 3D colonoscopy (Experimental): Use 3D machine to generate the 3D image
  Interventions: Device: 3D device
- 2D colonoscopy (No Intervention): Traditional colonoscopy

INTERVENTIONS:
Device: 3D device — Use 3D machine to generate the 3D image
  Arms: 3D colonoscopy

SUMMARY:
Background:

Adenoma detection rate is one of the most quality indicator: an accumulating body of evidence has shown that detection and resection of pre-cancerous adenoma by colonoscopy could effectively prevent colorectal cancer (CRC) and its related mortality1,2. Among various colonoscopy quality indicators, such as cecal intubation rate, withdrawal time, and adenoma detection rate (ADR), ADR is the most important one and most closely associated with the subsequent risk of CRC3,4. A recent study further demonstrated the improvement of ADR could reduce subsequent risk of CRC5.

Equipment and technique to improve ADR: To be noted, among all colorectal neoplasm, non-polypoid lesions, such as flat or depressed lesions, carries higher likelihood to be overlooked during conventional colonoscopy and these overlooked lesions were the main etiology of post-colonoscopy colorectal cancer (PCCRC)6. Nowadays, several colonoscopy technologies had been developed to enhance the detection of colorectal adenoma such as using digital or dye-spray chromoendoscopy7 or add-on device such as Cap/Endocuff/third eye/FUSE-assisted endoscopy8. Among them, some had showed the potential to enhance the detection of non-polypoid lesion, for example, the next-generation NBI9 or iSCAN10.

Application of 3D endoscopy on GI disease: 3D endoscopy is a new technology that using image processing technique to offer more information on tissue depth in comparison with conventional 2D endoscopy. The utility of 3D endoscopy on GI tract was mainly from upper GI tract and it was proved to enhance the diagnostic accuracy on superficial gastric tumors11 and shortened the procedure time during performing gastric endoscopic submucosal dissection (ESD)12. However, few is known that whether 3D colonoscopy could enhance the ADR, especially for non-polypoid lesion detection, during colonoscopy examination.

Positive fecal immunochemical test(FIT) group Among subjects who receive colonoscopy examination, higher advanced adenoma or invasive caners were found in FIT positive group. However, still about half of positive FIT subjects who received colonoscopy exam, have negative colonoscopy result. Non polypoid lesions could be overlooked during the colonoscopy. Therefore, we tried to use this prospective, multicenter, randomized control study to demonstrate the efficacy of 3D colonoscopy on adenoma detection in comparison with conventional 2D colonoscopy in this kind of high risk group.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are 40 years of older
* Subjects who have positive fecal immunochemical test

Exclusion Criteria:

* Contraindication for colonoscopy
* Subjects with familiar or hereditary polyposis
* Subjects with history of colectomy
* Inadequate bowel cleansing level
* Subjects with inflammatory bowel disease

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Adenoma detection rate | 30 minutes

SECONDARY OUTCOMES:
Flat-ADR | 30 minutes
  detection rate of flat adenoma
Proximal ADR | 30 minutes
  detection rate of adenoma at proximal colon
SSLDR | 30 minutes
  detection rate of sessile serrated lesion
AADR | 30 minutes
  detection rate of advanced adenoma
Polyp detection rate | 30 minutes
adenoma number per colonoscopy, | 30 minutes
polyp number per colonoscopy, | 30 minutes

CONTACTS AND LOCATIONS:
Locations (3):
- Taiwan (3):
  - National Taiwan University Cancer Center, Taipei, Taiwan
  - National Taiwan University Hospital, Taipei, Taiwan
  - National Taiwan University Hospital, Hsinchu Branch, Taoyuan District, Taiwan